CLINICAL TRIAL: NCT03411876
Title: Effects of an Oxymizer Pendant Cannula Versus a Conventional Nasal Cannula During Endurance Shuttle Walk Test (ESWT) in Hypoxemic Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Effects of Oxymizer Pendant Cannula Versus Conventional Nasal Cannula During Endurance Shuttle Walk Tests in Hypoxemic Patients With Idiopathic Pulmonary Fibrosis
Acronym: IPF/Oxymizer2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Kenn (Other)
Collaborators: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Sponsor-Investigator, Klaus Kenn, Prof. Dr. med., Schön Klinik Berchtesgadener Land
Organization: Schön Klinik Berchtesgadener Land (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IPF Oxymizer study II
Record Dates: First submitted 2018-01-18; First posted 2018-01-26 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Hypoxemia
Keywords: IPF; Oxymizer; oxygen conserving device; pulmonary disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypoxia; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- First ESWT with Oxymizer, second ESWT with CNC (Experimental): Patients in this study arm first perform the first endurance shuttle walk test (ESWT) with the Oxymizer and the second ESWT with a conventional nasal cannula (CNC).
  Interventions: Device: Oxymizer® pendant nasal cannula; Device: conventional nasal cannula
- First ESWT with CNC, second ESWT with Oxymizer (Experimental): Patients in this study arm first perform the first endurance shuttle walk test (ESWT) with the CNC and the second ESWT with the Oxymizer.
  Interventions: Device: Oxymizer® pendant nasal cannula; Device: conventional nasal cannula

INTERVENTIONS:
Device: Oxymizer® pendant nasal cannula — Supplemental oxygen is provided by an Oxymizer pendant nasal cannula.
Device: conventional nasal cannula — Supplemental oxygen is provided by a conventional nasal cannula.

SUMMARY:
Aim of this study is to investigate the effects of an Oxymizer pendant nasal cannula in hypoxemic patients with idiopathic pulmonary fibrosis during walking.

DETAILED DESCRIPTION:
Patients will be recruited during an inpatient pulmonary rehabilitation program. They will perform three shuttle walk tests on three consecutive days (see below). While performing those tests, the patient's prescribed oxygen flow rate is applicated either through the conventional nasal cannula (CNC) or the Oxymizer.On the first day, patients perform an incremental shuttle walk test to determine maximum walking speed using a conventional nasal cannula.

On two consecutive days, patients will perform two endurance shuttle walk tests at 85% of the maximum incremental shuttle walk test speed. Supplemental oxygen will be provided via nasal cannula at the prescribed oxygen flow rate. Patients will be randomly assigned to perform one test with the Oxymizer and the other one with a conventional nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* firmed diagnosis of idiopathic pulmonary fibrosis
* indication for supplemental oxygen therapy during exercise
* referred to an inpatient rehabilitation program at the Schön Klinik Berchtesgadener Land

Exclusion Criteria:

* cardiovascular diseases that influence the patient's physical performance
* orthopedic comorbidities that prevent the patient from performing an incremental or endurance shuttle walk test
* carbon dioxide pressure above 45 mmHg at rest and ambient air

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Endurance shuttle walk test distance | at baseline, at isotime of endurance shuttle walk test and at the end (maximum 20 min) of endurance shuttle walk test
  Distance patients walk during an endurance shuttle walk test

SECONDARY OUTCOMES:
oxygen saturation | at baseline, at isotime of endurance shuttle walk test and at the end (maximum 20 min) of endurance shuttle walk test
  measured by Sentec Digital Monitoring System
heart rate | at baseline, at isotime of endurance shuttle walk test and at the end (maximum 20 min) of endurance shuttle walk test
  measured by Sentec Digital Monitoring System
breathing frequency | at baseline, at isotime of endurance shuttle walk test and at the end (maximal 20 min) of endurance shuttle walk test
  measured by NoxT3 device
carbon dioxide pressure | at baseline, at isotime of endurance shuttle walk test and at the end (maximum 20 min) of endurance shuttle walk test
  transcutaneously carbon dioxide pressure measured by Sentec Digital Monitoring System
time to desaturation | From beginning of endurance shuttle walk test until the oxygen saturation reaches defined thresholds, or ESWT reaches maximum time frame of 20 minutes
  time (seconds) is measured until oxygen saturation drops below 90% or 85 % respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: No